CLINICAL TRIAL: NCT06241326
Title: A Real-world Study of Immunotherapy-based Combination Therapies in Chinese Patients With Hepatocellular Carcinoma
Brief Title: Immunotherapy for Hepatocellular Carcinoma
Acronym: IFHC
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-SR-876
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Hepatocellular Carcinoma; Immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- retrospective cohort: The patients in the retrospective cohort are hepatocellular carcinoma patients who have been previously treated with immunotherapy-based combination regimens. It is anticipated that approximately 10,000 cases will be included.
  Interventions: Other: Immunotherapy-based Combination Therapies
- prospective cohort: The patients included in the prospective cohort are hepatocellular carcinoma patients who are being evaluated by researchers to determine the potential benefits of undergoing immunotherapy-based combination treatment regimens. It is anticipated that approximately 1,000 cases will be enrolled.
  Interventions: Other: Immunotherapy-based Combination Therapies

INTERVENTIONS:
Other: Immunotherapy-based Combination Therapies — immunotherapy-based combination therapies in Chinese HCC patients within the practical context of real-world conditions

SUMMARY:
This study is an observational real-world research conducted on Chinese hepatocellular carcinoma (HCC) patients. Its primary objective is to evaluate the safety and efficacy of immunotherapy-based combination therapies in Chinese HCC patients within the practical context of real-world conditions.

DETAILED DESCRIPTION:
Hepatocellular carcinoma exhibits a significantly elevated incidence and mortality rate in China. Despite the Chinese population representing a mere 18.4% of the global population, the annual incidence of new liver cancer cases reaches a staggering 466,000 (55.4% of the global total), with 422,000 deaths (53.9% of the global total). Immunotherapy, particularly the implementation of immunotherapy-based combination treatment regimens, holds substantial therapeutic value in the management of hepatocellular carcinoma (HCC), leading to notable breakthroughs and advancements in the comprehensive treatment of liver cancer. The aim of this study is to evaluate the safety and efficacy of immunotherapy-based combination treatment regimens in Chinese hepatocellular carcinoma (HCC) patients under real-world clinical conditions. By collecting and analyzing data on the etiology, clinical characteristics, treatment modalities, and treatment outcomes of HCC patients receiving immunotherapy-based combination treatments in the clinical healthcare setting, the study seeks to provide valuable information regarding treatment patterns and effectiveness for hepatocellular carcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged after 18 years (18 is included).
2. Hepatocellular carcinoma diagnosed by pathology or imaging.
3. Patients assessed by researchers as potentially benefiting from receiving immunotherapy-based combination regimens.
4. For participants who have previously received treatment according to this protocol, a comprehensive pre-treatment assessment is required, including demographic information, tumor history, medical history, and baseline imaging examinations.
5. Patients voluntarily enroll in this study.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Other conditions regimented at investigators' discretion.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chinese hepatocellular carcinoma (HCC) patients
Sampling Method: Non-Probability Sample
Enrollment: 11000 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 24 months
  All adverse events during the course of the study treatment.

SECONDARY OUTCOMES:
Progression free survival | 24 months
  From date of admission until the date of first documented progression in the real-world setting or date of death from any cause, whichever came first, assessed up to 24 months.
Disease control rate | 24 months
  The percentage of subjects achieving complete response, partial response, or disease stability in a real-world clinical setting.
Objective response rate | 24 months
  The percentage of subjects achieving complete or partial response in a real-world clinical setting.
Duration of response | 24 months
  The time from the first documentation of objective response to the first assessment of progression in the real-world setting.
Overall survival | 24 months
  From date of admission until the date of death from any cause, assessed up to 24 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided